CLINICAL TRIAL: NCT06467201
Title: An Open-label, Sequential Dosing, Single Ascending Dose (SAD) Study to Determine the Safety, Tolerability, and Pharmacokinetic Profile of AMN1126 in Healthy Human Post-Menopausal Female Volunteers
Brief Title: SAD Study to Evaluate Safety, Tolerability, and Pharmacokinetic Profile of AMN1126 in Healthy Post-Menopausal Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shivanka Research, LLC (Industry)
Collaborators: Amneal Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CE-24-02
Record Dates: First submitted 2024-06-08; First posted 2024-06-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy Postmenopausal Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KSHN001126 150mg (Experimental): Low Dose
  Interventions: Drug: KSHN001126 150mg
- KSHN001126 300mg (Experimental): Mid Dose
  Interventions: Drug: KSHN001126 300mg
- KSHN001126 600mg (Experimental): High Dose
  Interventions: Drug: KSHN001126 600mg

INTERVENTIONS:
Drug: KSHN001126 150mg — 6 subjects will receive single oral dose of 150mg
  Arms: KSHN001126 150mg
Drug: KSHN001126 300mg — 6 subjects will receive single oral dose of 300mg
  Arms: KSHN001126 300mg
Drug: KSHN001126 600mg — 6 subjects will receive single oral dose of 600mg
  Arms: KSHN001126 600mg

SUMMARY:
This is an Open-label, Sequential dosing, Single Ascending Dose (SAD) Study to Determine the Safety, Tolerability, and Pharmacokinetic (PK) Profile of KSHN001126 in Healthy Human Post-Menopausal Female Volunteers. The primary objective of the study is to evaluate the safety and tolerability of increasing single doses of KSHN001126 while the secondary objective is to evaluate the plasma PK profile of KSHN001126 and its metabolites (KSHN001167, KSHN001168 and Fulvestrant) following ascending single oral doses of KSHN001126.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written Informed Consent and communicate with the investigator and comprehend study-related procedures.
2. Healthy, postmenopausal females aged 45 to 60 years old (inclusive), as determined by medical history and physical examination.
3. Body Mass Index at screening between 18 and 30 kg/m2, inclusive.
4. Post-menopausal females (Menopause is defined as the female is either 12 months off menstrual period after the age of 50 years, or 12 months off menstrual period after the age of 40 years and Follicle Stimulating Hormone (FSH) > 40 mIU/mL. Amenorrhea should not be due to lactation).
5. In good general health with no clinically significant illness seen on physical examination or ongoing medical history, as determined by the Investigator.
6. Documented 12-lead ECG with no clinically significant abnormalities (with QTc interval between 360 to 440 msec), as determined by the Investigator in screening or Day 0.
7. No clinically significant abnormalities in screening or Day 0 laboratory tests, as determined by the Investigator (Creatinine clearance should be ≥ 90 mL/min and Blood Urea Nitrogen / AST / ALT / Alkaline phosphatase / Total and direct bilirubin should be < upper limit of normal).
8. Female participants must have a negative serum pregnancy (β-HCG) test at screening and a negative urine pregnancy test at Day 0 prior to dosing. Female participants must also be non-lactating.
9. The participant is available to volunteer for the entire study duration and is willing to adhere to all protocol requirements.
10. The participant has vital signs at screening, and at check-in within the following ranges:

    * Blood Pressure:

      * Systolic: (100- 140 mmHg
      * Diastolic: (60-90) mmHg
    * Body Temperature: (36.1 - 37.8) ºC, Pulse rate: 60 to 100 b/m. Respiratory rate: 12 to 20 bpm
11. Participants with normal findings as determined by gynecological examination and USG Pelvis.
12. With a normal or clinically acceptable mammogram
13. With a normal or clinically acceptable PAP smear test
14. Have a normal chest X-ray (P. A. view).
15. Participant negative for hepatitis B-surface antigen, hepatitis C and Human Immunodeficiency Virus (HIV)
16. Participants who are generally healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring
17. Adequate venous access and can able to give required blood samples.

Exclusion Criteria:

1. The participant is surgically induced postmenopausal female.
2. Pregnant or lactating female participant.
3. Any history of clinically significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, chronic hepatic disease or any other disease which in the judgment of the Investigator would interfere with the study or confound the study results.
4. History of allergy or major allergic reaction considered to be clinically significant by the Investigator.
5. Receiving or has received any investigational drug within the 30 days before receiving KSHN001126.
6. History or presence of low platelet count, bleeding issues or family history of bleeding disorders.
7. Participant has a history of hypersensitivity to heparin as checked at screening.
8. The participant has known allergy to the drug under investigation, or to any ingredient in the preparation
9. The participant has an evidence of antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of the consent to participation in the study or limit the ability to comply with the protocol requirements.
10. Donated blood within 60 days of screening or otherwise experienced blood loss of >250 mL within the same period.
11. Intending to begin new concomitant drug therapy or over-the-counter medication anytime from screening to the time of administration of study drug.
12. Received or intending to receive a vaccination in the two weeks prior to dosing, or anytime during study participation.
13. Received treatment with a drug that has not received regulatory approval for an indication during the 60 days preceding study enrollment.
14. History of drug and/or alcohol dependence within past 12 months, and/or positive results on drug of abuse or alcohol tests.
15. The participant is a smoker (smoker is defined as reporting tobacco use in the previous 3 months and/or has urine cotinine level equal or more than 500 ng/ml)
16. Has taken any regular, prescribed, or over-the-counter medication with the exception of acetaminophen (maximum 2 g/day) or multi- vitamins in the 2 weeks prior to dosing (other medication may only be taken with the specific approval of the Investigator in consultation with the Medical Monitor).
17. The participant with history of consuming alcohol or caffeine or related xanthine containing foods or beverages such as caffeine in tea, coffee, chocolates, cola and pepsi for 48 hours prior to dosing.
18. The participant has consumed grapefruit-containing beverages and foods 7 days prior to dosing.
19. Malignancy within the last 5 years, with the exception of successfully treated basal cell carcinoma and carcinoma in situ uteri.
20. The participant has prior history of hormonal replacement therapy.
21. The participant has any estrogen- dependent conditions including breast cancer.
22. Any condition that, in the opinion of the investigator, might interfere with study objectives.
23. The participant has a history of osteoporosis or any disease affecting bone or steroid metabolism.
24. Intolerance to/ fear of venipuncture, needles, or blood draws

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Type, incidence, severity, seriousness, and relatedness of Adverse Events (AEs) | Upto Day 15 after dosing
  Adverse events reported after dosing will be evaluated
Number of participants with abnormal laboratory tests results | Upto Day 15 after dosing
  Laboratory abnormalities after dosing will be evaluated
Number of participants with abnormal vital signs | Upto Day 15 after dosing
Number of participants with abnormal Electrocardiogram readings | Upto Day 15 after dosing
  Impact on QTc interval will be evaluated

SECONDARY OUTCOMES:
Evaluate the Peak Plasma Concentration (Cmax) of KSHN001126 and its metabolites (KSHN001167, KSHN001168 and Fulvestrant) following ascending single oral doses of KSHN001126 | 72 hours after dosing
Evaluate the Area under the plasma concentration versus time curve (AUC) of KSHN001126 and its metabolites (KSHN001167, KSHN001168 and Fulvestrant) following ascending single oral doses of KSHN001126 | 72 hours after dosing
Evaluate the Time to maximum concentration (Tmax) of KSHN001126 and its metabolites (KSHN001167, KSHN001168 and Fulvestrant) following ascending single oral doses of KSHN001126 | 72 hours after dosing
Evaluate the half life (T1/2) of KSHN001126 and its metabolites (KSHN001167, KSHN001168 and Fulvestrant) following ascending single oral doses of KSHN001126 | 72 hours after dosing

CONTACTS AND LOCATIONS:
Locations (2):
- Advanced Pharma CR, Miami, Florida, United States
- Health1 Superspeciality Hospital, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No